CLINICAL TRIAL: NCT04576988
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Compare the Efficacy and Safety of Sotatercept Versus Placebo When Added to Background Pulmonary Arterial Hypertension (PAH) Therapy for the Treatment of PAH
Brief Title: A Study of Sotatercept for the Treatment of Pulmonary Arterial Hypertension (MK-7962-003/A011-11)(STELLAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7962-003; 7962-003 (Other: MSD); 2020-004142-11 (EudraCT Number)
Record Dates: First submitted 2020-09-28; First posted 2020-10-06 (Actual); Results first posted 2023-08-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — ACE-011

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two treatment arms to receive either sotatercept (0.7 mg/kg) by subcutaneous administration once every 3 weeks, or placebo. All participants will be on concurrent, stable background PAH therapy. Randomization will be stratified by baseline WHO Functional Class (Class II or III) and by background PAH therapy (mono/double or triple therapy)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study participants, care providers. Investigators and outcomes assessor will be masked to the study intervention until the final participant completes the 24-week efficacy assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sotatercept plus background PAH therapy (Experimental): Sotatercept at a starting dose of 0.3 mg/kg with a target dose of 0.7 mg/kg administered subcutaneously (SC) every 21 days plus background PAH therapy
  Interventions: Biological: Sotatercept; Drug: Background PAH Therapy
- Placebo plus background PAH therapy (Placebo Comparator): Placebo administered (SC) every 21 days plus background PAH therapy
  Interventions: Drug: Placebo; Drug: Background PAH Therapy

INTERVENTIONS:
Biological: Sotatercept — Sotatercept at a starting dose of 0.3 mg/kg with a target dose of 0.7 mg/kg administered subcutaneously (SC) every 21 days plus background PAH therapy.
  Other Names: MK-7962; ACE-011
  Arms: Sotatercept plus background PAH therapy
Drug: Placebo — Placebo administered subcutaneously (SC) every 21 days plus background PAH therapy.
  Arms: Placebo plus background PAH therapy
Drug: Background PAH Therapy — Background PAH therapy may consist of the following drug classes: an endothelin-receptor antagonist (ERA), a phosphodiesterase 5 (PDE5) inhibitor, a soluble guanylate cyclase stimulator, and/or a prostacyclin analogue or receptor agonist.

SUMMARY:
The objectives of this study are to evaluate the efficacy and safety of sotatercept (MK-7962) treatment (plus background pulmonary arterial hypertension (PAH) therapy) versus placebo (plus background PAH therapy) at 24 weeks in adults with PAH. The primary hypothesis of the study is that the participants receiving sotatercept will have improved 6-minute walk distance (6MWD) at 24 weeks compared to participants receiving placebo.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, multicenter, parallel-group study in subjects with symptomatic PAH who present with idiopathic or heritable PAH, PAH associated with connective tissue diseases (CTD), drug or toxin induced, post shunt correction PAH, or PAH presenting at least 1 year following the correction of congenital heart defects (CHDs), and currently on background PAH therapy.

The primary efficacy endpoint of the study is exercise capacity, as measured by the 6-minute walk distance (6MWD) measured at 24 week following initiation of treatment.

Study duration will be approximately 2 years. A stratified Wilcoxon test will be used for analysis of the primary endpoint, with appropriate imputation for missing data, as detailed in the Statistical Analysis Plan. An unblinded, external, independent Data Monitoring Committee (DMC) will monitor participant safety throughout the course of the study. Participants completing this study will be eligible to receive sotatercept in a separate, open-label extension study.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years
* Documented diagnostic right heart catheterization (RHC) at any time prior to screening confirming the diagnosis of World Health Organization (WHO) pulmonary arterial hypertension (PAH) Group 1 in any of the following subtypes:

  * Idiopathic PAH
  * Heritable PAH
  * Drug/toxin-induced PAH
  * PAH associated with connective tissue disease
  * PAH associated with simple, congenital systemic to pulmonary shunts at least 1 year following repair
* Symptomatic PAH classified as WHO Functional Class (FC) II or III
* Baseline RHC performed during the Screening Period documenting a minimum pulmonary vascular resistance (PVR) of ≥ 5 Wood units (WU) and a pulmonary capillary wedge pressure (PCWP) or left ventricular end-diastolic pressure of ≤ 15 mmHg.
* On stable doses of background PAH therapy and diuretics (i.e., patient-specific dose goal for each therapy already achieved) for at least 90 days prior to screening; for infusion prostacyclins, dose adjustment within 10% of optimal dose is allowed per medical practice

  * Background PAH therapy refers to approved PAH-specific medications and may consist of monotherapy or combination therapy with ERA, PDE5 inhibitors, soluble guanylate cyclase stimulators, and/or prostacyclin analogues or receptor agonists. Background PAH therapy should be stable at least 90 days prior to screening and remain stable throughout the study
  * Stable diuretic therapy is defined as no addition of a new diuretic and no switching of a pre-existent oral diuretic to parenteral administration; however, dose adjustments (up or down) in pre-existent oral diuretics are acceptable
* 6-Minute Walk Distance (6MWD) ≥ 150 and ≤ 500 m repeated twice at screening (measured at least 4 hours apart, but no longer than 1 week), and both values are within 15% of each other (calculated from the highest value)
* Females of childbearing potential must:

  * Have 2 negative urine or serum pregnancy tests as verified by the investigator prior to starting study therapy; she must agree to ongoing urine or serum pregnancy testing during the study and until 8 weeks after the last dose of the study drug
  * If sexually active, have used, and agree to use, highly effective contraception without interruption, for at least 28 days prior to starting the investigational product, during the study (including dose interruptions), and for 16 weeks (112 days) after discontinuation of study treatment
  * Refrain from breastfeeding a child or donating blood, eggs, or ovum for the duration of the study and for at least 16 weeks (112 days) after the last dose of study treatment
  * Male participants must:
  * Agree to use a condom, defined as a male latex condom or nonlatex condom NOT made out of natural (animal) membrane (e.g., polyurethane), during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 16 weeks (112 days) following investigational product discontinuation, even if he has undergone a successful vasectomy
  * Refrain from donating blood or sperm for the duration of the study and for 16 weeks (112 days) after the last dose of study treatment
  * Ability to adhere to study visit schedule and understand and comply with all protocol requirements
  * Ability to understand and provide written informed consent

Key Exclusion Criteria:

* Diagnosis of pulmonary hypertension WHO Groups 2, 3, 4, or 5
* Diagnosis of the following PAH Group 1 subtypes: human immunodeficiency virus (HIV)-associated PAH and PAH associated with portal hypertension. Exclusions in PAH Group I should also include schistosomiasis associate PAH and pulmonary veno occlusive disease
* Hemoglobin (Hgb) at screening above gender-specific upper limit of normal (ULN), per local laboratory test
* Baseline platelet count < 50,000/mm^3 (< 50.0 x 109/L) at screening
* Uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure > 160 mmHg or sitting diastolic blood pressure > 100 mmHg during screening visit after a period of rest
* Baseline systolic blood pressure < 90 mmHg at screening
* Pregnant or breastfeeding women
* Any of the following clinical laboratory values at the screening visit:

  * Estimated glomerular filtration rate (eGFR) < 30 mL/min/m2 (as defined by the Modification of Diet in Renal Disease [MDRD] equation)
  * Serum alanine aminotransferase, aspartate aminotransferase, or total bilirubin levels > 3 × ULN (bilirubin criterion waived if there is a documented history of Gilbert's syndrome)
* Currently enrolled in or have completed any other investigational product study within 30 days for small molecule drugs or within 5 half-lives for biologics prior to the date of signed informed consent
* Prior exposure to sotatercept (ACE-011) or luspatercept (ACE 536) and/or excipients or known allergic reaction to either one
* History of full pneumonectomy
* Pulmonary function test (PFT) values of forced vital capacity (FVC) < 60% predicted at the screening visit or within 6 months prior to the screening visit. If PFT is not available, a chest CT scan showing more than mild interstitial lung disease (ILD) at the screening visit or 1 year prior to it
* Initiation of an exercise program for cardiopulmonary rehabilitation within 90 days prior to the screening visit or planned initiation during the study (participants who are stable in the maintenance phase of a program and who will continue for the duration of the study are eligible)
* History of more than mild obstructive sleep apnea that is untreated
* Known history of portal hypertension or chronic liver disease, including hepatitis B and/or hepatitis C (with evidence of recent infection and/or active virus replication), defined as mild to severe hepatic impairment (Child-Pugh Class A-C)
* History of restrictive, constrictive or congestive cardiomyopathy
* History of atrial septostomy within 180 days prior to the screening visit
* Electrocardiogram (ECG) with Fridericia's corrected QT interval (QTcF) > 500 ms during the screening period
* Personal or family history of long QT syndrome (LQTS) or sudden cardiac death
* Left ventricular ejection fraction < 45% on historical echocardiogram within 6 months prior to the screening visit
* Any symptomatic coronary disease events (prior myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft surgery, or cardiac anginal chest pain) within 6 months prior to the screening visit. Note: Anginal pain can be ignored as an exclusion criterion if coronary angiography shows no obstructions
* Cerebrovascular accident within 3 months prior to the screening visit
* Acutely decompensated heart failure within 30 days prior to the screening visit, as per investigator assessment
* Significant (≥ 2+ regurgitation) mitral regurgitation or aortic regurgitation valvular disease
* Received intravenous inotropes (e.g., dobutamine, dopamine, norepinephrine, vasopressin) within 30 days prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (120):
- United States (39):
  - Arizona Pulmonary Specialists (Site 1010), Phoenix, Arizona
  - Pulmonary Associates, PA (Site 1008), Phoenix, Arizona
  - University of Arizona (Site 1006), Tucson, Arizona
  - University of California San Diego Medical Center (Site 1002), San Diego, California
  - University of California - Davis Medical Center (Site 1064), Sherman Oaks, California
  - Stanford University Medical Center (Site 1024), Stanford, California
  - Harbor UCLA Medical Center (Site 1028), Torrance, California
  - University of Colorado Hospital (Site 1013), Aurora, Colorado
  - The George Washington University Medical Faculty Associates (Site 1025), Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville (Site 1045), Jacksonville, Florida
  - University of South Florida (Site 1043), Tampa, Florida
  - The Emory Clinic (Site 1030), Atlanta, Georgia
  - Norton Pulmonary Specialists (Site 1066), Louisville, Kentucky
  - Tufts Medical Center - PPDS (Site 1012), Boston, Massachusetts
  - Brigham and Women's Hospital (Site 1014), Boston, Massachusetts
  - University of Michigan (Site 1011), Ann Arbor, Michigan
  - University of Minnesota (Site 1062), Minneapolis, Minnesota
  - Mayo Clinic (Site 1023), Rochester, Minnesota
  - University of Kansas Medical Center (Site 1020), Kansas City, Missouri
  - Washington University School of Medicine (Site 1022), St Louis, Missouri
  - Nebraska Medical Center (Site 1053), Omaha, Nebraska
  - Renown Institute for Heart & Vascular Health (Site 1055), Reno, Nevada
  - New York Presbyterian Hospital (Site 1046), New York, New York
  - Duke University Medical Center (Site 1026), Durham, North Carolina
  - University of Cincinnati Medical Center (Site 1035), Cincinnati, Ohio
  - The Carl and Edyth Lindner Center for Research and Education at the Christ Hospital (Site 1001), Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center (Site 1005), Cleveland, Ohio
  - The Ohio State University Wexner Medical Center (Site 1032), Columbus, Ohio
  - Oregon Health and Science University (Site 1054), Portland, Oregon
  - University of Pennsylvania (Site 1047), Philadelphia, Pennsylvania
  - UPMC Presbyterian. UPMC Presbyterian Hospital (Site 1059), Pittsburgh, Pennsylvania
  - Rhode Island Hospital (Site 1033), Providence, Rhode Island
  - Medical University of South Carolina - PPDS (Site 1003), Charleston, South Carolina
  - Statcare Pulmonary Consultants - Knoxville (Site 1031), Knoxville, Tennessee
  - Vanderbilt University Medical Center (Site 1027), Nashville, Tennessee
  - CHI St. Luke's Health Baylor College of Medicine Medical Center (Site 1044), Houston, Texas
  - Houston Methodist Hospital (Site 1009), Houston, Texas
  - University of Utah - PPDS (Site 1049), Salt Lake City, Utah
  - University of Washington Medical Center - Montlake (Site 1067), Seattle, Washington
- Argentina (5):
  - Hospital Universitario Austral ( Site 1901), Pilar, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes ( Site 1903), Quilmes, Buenos Aires
  - Centro Medico Dra De Salvo ( Site 1904), Buenos Aires, Buenos Aires F.D.
  - Sanatorio Parque ( Site 1905), Rosario, Santa Fe Province
  - Hospital Provincial Dr. Jose M. Cullen ( Site 1902), Santa Fe
- Australia (6):
  - Royal Prince Alfred Hospital ( Site 1106), Camperdown, New South Wales
  - Saint Vincents Hospital Sydney ( Site 1102), Darlinghurst, New South Wales
  - John Hunter Hospital ( Site 1101), New Lambton, New South Wales
  - Westmead Hospital ( Site 1105), Westmead, New South Wales
  - Prince Charles Hospital ( Site 1104), Chermside, Queensland
  - The Alfred Hospital ( Site 1110), Melbourne, Victoria
- Belgium (2):
  - Hopital Erasme ( Site 1402), Brussels, Bruxelles-Capitale, Region de
  - U.Z.-Gasthuisberg ( Site 1401), Leuven, Vlaams-Brabant
- Brazil (3):
  - Irmandade da Santa Casa de Misericordia de Porto Alegre ( Site 1805), Porto Alegre, Rio Grande do Sul
  - Hospital Dia do Pulmao ( Site 1802), Blumenau, Santa Catarina
  - Instituto do Coracao - HC FMUSP ( Site 1803), São Paulo
- Canada (3):
  - University Of Alberta Hospital ( Site 2101), Edmonton, Alberta
  - University of Ottawa Heart Institute ( Site 2104), Ottawa, Ontario
  - Jewish General Hospital ( Site 2103), Montreal, Quebec
- Czechia (3):
  - Fakultni Nemocnice Olomouc ( Site 2203), Olomouc, Olomoucký kraj
  - Institut Klinicke a Experimentalni Mediciny ( Site 2202), Prague, Praha 4
  - Vseobecna fakultni nemocnice v Praze ( Site 2201_, Prague, Praha, Hlavni Mesto
- France (13):
  - Hopital Pasteur (Site 1311), Nice, Alpes-Maritimes
  - Hopitaux Universitaires de Strasbourg ( Site 1307), Strasbourg, Bas-Rhin
  - CHRU Brest - Hopital Cavale Blanche (Site 1314), Brest, Finistere
  - Groupe Hospitalier Sud ( Site 1312), Pessac, Gironde
  - CHU de Toulouse - Hopital Larrey ( Site 1315), Toulouse, Haute-Garonne
  - Hopital Arnaud de Villeneuve ( Site 1301), Montpellier, Herault
  - CHU de Grenoble - Hopital Michallon ( Site 1303), Grenoble, Isere
  - CHU Nantes - Hopital Laennec (Site 1309), Nantes, Loire-Atlantique
  - CHU Angers (Site 1313), Angers, Maine-et-Loire
  - C.H.U. de Nancy. Hopital de Brabois Adultes ( Site 1308), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHRU Lille ( Site 1306), Lille, Nord
  - Centre Hospitalier Universitaire de Saint-Etienne ( Site 1302), Saint-Priest-en-Jarez, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Bicetre ( Site 1304), Le Kremlin-Bicêtre, Val-de-Marne
- Germany (9):
  - Thoraxklinik-Heidelberg gGmbH (Site 1509), Heidelberg, Baden-Wurttemberg
  - Krankenhaus Neuwittelsbach (Site 1510), Munich, Bavaria
  - Universitaetsklinik Regensburg (Site 1503), Regensburg, Bavaria
  - Universitaetsklinikum Giessen und Marburg GmbH ( Site 1512), Giessen, Hesse
  - Medizinische Hochschule Hannover (Site 1505), Hanover, Lower Saxony
  - Uniklinik Köln, Institut für Kliniche Chemie ( Site 1511), Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus der TU Dresden (Site 1501), Dresden, Saxony
  - Universitätsklinikum Halle (Site 1502), Halle, Saxony-Anhalt
  - DRK Kliniken Berlin Westend ( Site 1507), Berlin
- Israel (4):
  - Lady Davis Carmel Medical Center (Site 1705), Haifa
  - Meir Medical Center (Site 1707), Kfar Saba
  - Rabin Medical Center (Site 1703), Petah Tikva
  - Sheba Medical Center (Site 1701), Tel Litwinsky
- Universita "La Sapienza" Policlinico Umberto I (Site 2402), Roma, Italy
- Mexico (3):
  - CIMAB SA de CV (Site 2502), Torreón, Coahuila
  - Unidad de Investigacion Clinica en Medicina, S.C. (Site 2505), Monterrey, Nuevo León
  - Operadora de Hospitales Angeles. S.A. de C.V. -Sucursal Lomas (Site 2501), Huixquilucan
- Netherlands (2):
  - Maastricht University Medical Center (Site 2603), Maastricht, Limburg
  - VU Medisch Centrum (Site 2601), Amsterdam, North Holland
- New Zealand (3):
  - University of Otago, Wellington (Site 2701), Christchurch, Canterbury
  - Waikato District Health Board (Site 2702), Hamilton, Waikato Region
  - Greenlane Clinical Centre (Site 2703), Auckland
- Poland (3):
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II (Site 2801), Krakow, Lesser Poland Voivodeship
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina (Site 2802), Otwock, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku (Site 2803), Bialystok, Podlaskie Voivodeship
- Serbia (3):
  - Clinical Center of Serbia (Site 2901), Belgrade, Beograd
  - Institute of Cardiovascular Diseases Dedinje (Site 2903), Belgrade, Beograd
  - University Clinical Center Nis (Site 2904), Niš, Nisavski Okrug
- South Korea (3):
  - Gachon University Gil Medical Center (Site 3103), Incheon
  - Seoul National University Hospital (Site 3102), Seoul
  - Severance Hospital Yonsei University Health System - PPDS (Site 3101), Seoul
- Spain (7):
  - Hospital Universitario Marques de Valdecilla (Site 1601), Santander, Cantabria
  - Hospital Universitario Puerta de Hierro-Majadahonda (Site 1604), Majadahonda, Madrid
  - Hospital Universitari Vall d'Hebron (Site 1605), Barcelona
  - Hospital Clinic de Barcelona (Site 1602), Barcelona
  - Hospital Universitario Ramon y Cajal (Site 1609), Madrid
  - Hospital Universitario Marques de Valdecilla (Site 1603), Madrid
  - Hospital Clinico Universitario de Salamanca (Site 1608), Salamanca
- Sweden (2):
  - Akademiska Sjukhuset (Site 3204), Uppsala, Uppsala County
  - Sahlgrenska Universitets Sjukhuset (Site 3201), Gothenburg, Västra Götaland County
- Switzerland (2):
  - Hopitaux Universitaires de Geneve HUG (Site 3302), Thônex, Canton of Geneva
  - Universitaetsspital Zuerich (Site 3301), Zurich
- United Kingdom (4):
  - Golden Jubilee National Hospital (Site 1204), Glasgow, Glasgow City
  - Royal Free London NHS Foundation Trust (Site 1202), London, London, City of
  - Royal Brompton Hospital (Site 1206), London, London, City of
  - Imperial College Healthcare NHS Trust (Site 1203), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hoeper MM, Badesch DB, Ghofrani HA, Gibbs JSR, Gomberg-Maitland M, McLaughlin VV, Preston IR, Souza R, Waxman AB, Grunig E, Kopec G, Meyer G, Olsson KM, Rosenkranz S, Xu Y, Miller B, Fowler M, Butler J, Koglin J, de Oliveira Pena J, Humbert M; STELLAR Trial Investigators. Phase 3 Trial of Sotatercept for Treatment of Pulmonary Arterial Hypertension. N Engl J Med. 2023 Apr 20;388(16):1478-1490. doi: 10.1056/NEJMoa2213558. Epub 2023 Mar 6. PMID 36877098
- [Derived] Alsumali A, McLaughlin V, Chevure J, Klok R, Zhang W, Martinez EC, Pausch C, De Oliveira Pena J, van de Wetering G, Jootun M, Lautsch D, Hoeper MM. Long-Term Mortality and Morbidity Impact on Patients with Pulmonary Arterial Hypertension (PAH) If Access to Sotatercept Is Delayed: A Simulation Model. Adv Ther. 2025 Aug;42(8):3902-3921. doi: 10.1007/s12325-025-03241-4. Epub 2025 Jun 17. PMID 40526255
- [Derived] McLaughlin V, Alsumali A, Liu R, Klok R, Martinez EC, Nourhussein I, Bernotas D, Chevure J, Pausch C, De Oliveira Pena J, Lautsch D, Hoeper MM. Population Health Model Predicting the Long-Term Impact of Sotatercept on Morbidity and Mortality in Patients with Pulmonary Arterial Hypertension (PAH). Adv Ther. 2024 Jan;41(1):130-151. doi: 10.1007/s12325-023-02684-x. Epub 2023 Oct 18. PMID 37851297
- [Derived] Souza R, Badesch DB, Ghofrani HA, Gibbs JSR, Gomberg-Maitland M, McLaughlin VV, Preston IR, Waxman AB, Grunig E, Kopec G, Meyer G, Olsson KM, Rosenkranz S, Lin J, Johnson-Levonas AO, de Oliveira Pena J, Humbert M, Hoeper MM. Effects of sotatercept on haemodynamics and right heart function: analysis of the STELLAR trial. Eur Respir J. 2023 Sep 21;62(3):2301107. doi: 10.1183/13993003.01107-2023. Print 2023 Sep. PMID 37696565
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26050&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 324 randomized participants, 1 participant was randomized in error and did not receive study treatment and no data was collected. Hence, the results are presented on 323 participants.
Pre-assignment Details: Per protocol, not all participants from the double-blind placebo controlled (DBPC) period entered the long-term double blind (LTDB) period due to clinical worsening or consent withdrawal after DBPC period.
Groups:
- Sotatercept Plus Background PAH Therapy: Participants received a starting dose of sotatercept 0.3 mg/kg titrated up to 0.7mg/kg by subcutaneous (SC) injection every 21 days plus background PAH therapy during the double-blind placebo controlled (DBPC) period for up to approximately 24 weeks. After 24 weeks, participants received sotatercept dose titrated up to 0.7mg/kg SC injection every 21 days plus background PAH therapy during the long-term double blind (LTDB) period for up to approximately 72 weeks.
- Placebo Plus Background PAH Therapy: Participants received dose matched placebo by SC injection every 21 days plus background PAH therapy during the DBPC period for up to approximately 24 weeks and the LTDB period for up to approximately 72 weeks.
Period: Double Blind Placebo Controlled (DBPC)
Arm/Group | Sotatercept Plus Background PAH Therapy | Placebo Plus Background PAH Therapy
Started | 163 | 160
Treated | 163 | 160
Completed | 159 | 148
Not Completed | 4 | 12
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Death | 0 | 5
Not completed — Clinical worsening event | 0 | 2
Period: Long Term Double Blind (LTDB)
Arm/Group | Sotatercept Plus Background PAH Therapy | Placebo Plus Background PAH Therapy
Started | 159 | 142 (Not all participants from placebo plus background PAH arm in the DBPC period entered the LTDB period due to clinical worsening or consent withdrawal after DBPC period.)
Treated | 158 | 142
Completed | 155 | 136
Not Completed | 4 | 6
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Death | 2 | 1
Not completed — Sponsor decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Of the 324 participants randomized in the study, one participant was randomized in error in placebo plus background PAH therapy arm and no data was collected on this participant. Per protocol, this participant was excluded from the study analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sotatercept Plus Background PAH Therapy | Placebo Plus Background PAH Therapy | Total
Number analyzed (Participants) | 163 | 160 | 323
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.6 (14.09) | 48.3 (15.50) | 47.9 (14.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 127 | 256
  Male | 34 | 33 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 31 | 58
  Not Hispanic or Latino | 132 | 124 | 256
  Unknown or Not Reported | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 5 | 7
  White | 147 | 141 | 288
  More than one race | 7 | 4 | 11
  Unknown or Not Reported | 6 | 2 | 8
6-Minute Walk Distance (6MWD) at baseline [Mean (Standard Deviation); unit: meters] — The 6MWD is the distance walked in 6 minutes as a measure of functional capacity.
  meters | 397.6 (84.28) | 404.7 (80.59) | 401.1 (82.4)
World Health Organization (WHO) functional class (FC) II or III at baseline [Count of Participants; unit: Participants] — WHO FC was used to rate how ill a pulmonary arterial hypertension (PAH) participant was.
  Class II: Participants with PAH resulting in a slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity causes undue dyspnea or fatigue, chest pain, or near syncope.
  Class III: Participants with PAH resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes undue dyspnea or fatigue, chest pain, or near syncope
  Participants
    Class II | 79 | 78 | 157
    Class III | 84 | 82 | 166
Background PAH Therapy at Baseline [Count of Participants; unit: Participants] — Background PAH therapy refers to approved PAH-specific medications and may consist of monotherapy or combination therapy (double or triple therapy) with endothelin-receptor antagonist (ERA), a phosphodiesterase 5 (PDE5) inhibitors, soluble guanylate cyclase stimulators, and/or prostacyclin analogues or receptor agonists.
  Participants
    Monotherapy | 9 | 4 | 13
    Double therapy | 56 | 56 | 112
    Triple therapy | 98 | 100 | 198

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 6-Minute Walk Distance (6MWD) at Week 24
Description: The 6MWD was the distance walked in 6 minutes as a measure of functional capacity. This was assessed using the 6-minute walk test (6MWT). Per protocol, change from baseline in 6MWD at Week 24 was reported for DBPC period.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of study treatment and had a baseline value of 6MWD.
Measure: Median (Full Range); unit: meters
Groups:
- Sotatercept Plus Background PAH Therapy (DBPC Period): Participants received a starting dose of sotatercept 0.3 mg/kg titrated up to 0.7mg/kg by subcutaneous (SC) injection every 21 days plus background PAH therapy during the DBPC period for up to approximately 24 weeks.
- Placebo Plus Background PAH Therapy (DBPC Period): Participants received dose matched placebo by SC injection every 21 days plus background PAH therapy during the DBPC period for up to approximately 24 weeks.
Arm/Group | Sotatercept Plus Background PAH Therapy (DBPC Period) | Placebo Plus Background PAH Therapy (DBPC Period)
Number analyzed (Participants) | 163 | 160
meters | 34.4 [32.5 to 35.5] | 1.0 [-1.0 to 5.0]
Statistical Analysis 1: Comparison: Sotatercept Plus Background PAH Therapy (DBPC Period) vs Placebo Plus Background PAH Therapy (DBPC Period); Test type: Other; p < 0.001, Aligned Rank Stratified Wilcoxon (ARSW) — A 2-sided p-value was calculated using ARSW test with WHO FC II/III and background PAH therapy as strata; Participants who died were assigned the worst rank and who had missing data due to non-fatal clinical worsening event were assigned next worst-rank; Treatment difference = 40.8, 95% CI 2-sided [27.53 to 54.14] — Hodges-Lehmann location-shift estimate of the overall treatment difference with 95% confidence interval (CI) was reported

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a study participant administered a study drug, which did not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it was considered related to the study drug. Per protocol, the number of participants who reported an AE were reported for DBPC period.
Time Frame: Up to approximately 24 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept Plus Background PAH Therapy (DBPC Period) | Placebo Plus Background PAH Therapy (DBPC Period)
Number analyzed (Participants) | 163 | 160
Participants | 138 | 140

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a study participant administered a study drug, which did not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it was considered related to the study drug. Per protocol, the number of participants who discontinued study treatment due to an AE were reported for DBPC period.
Time Frame: Up to approximately 24 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept Plus Background PAH Therapy (DBPC Period) | Placebo Plus Background PAH Therapy (DBPC Period)
Number analyzed (Participants) | 163 | 160
Participants | 3 | 10

4. Secondary Outcome: Change From Baseline in the Percentage of Participants Achieving Multicomponent Improvement at Week 24
Description: Multicomponent Improvement was defined as consisting of all of the following: (a) Improvement in 6MWD (increase ≥30 meters) (b) Improvement in N-terminal pro b-type natriuretic peptide (NT-proBNP; decrease in NT-proBNP ≥30%) or maintenance/achievement of NT-proBNP level <300 ng/L (c) Improvement in World Health Organization (WHO) Functional Class (FC) or maintenance of WHO FC II. Per protocol, change from baseline in the percentage of participants achieving multicomponent improvement at Week 24 was reported for DBPC period.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of study treatment and who had a baseline measurement for the multicomponent improvement.
Measure: Number; unit: Percent change
Groups:
- Placebo Plus Background PAH Therapy (DBPC Period): Participants received dose matched placebo SC injection every 21 days plus background PAH therapy during the DBPC period for up to approximately 24 weeks.
Arm/Group | Sotatercept Plus Background PAH Therapy (DBPC Period) | Placebo Plus Background PAH Therapy (DBPC Period)
Number analyzed (Participants) | 162 | 159
Percent change | 38.9 | 10.1
Statistical Analysis 1: Comparison: Sotatercept Plus Background PAH Therapy (DBPC Period) vs Placebo Plus Background PAH Therapy (DBPC Period); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; A 2-sided p-value was calculated using Cochran-Mantel-Haenszel (CMH) method with WHO FC II/III and background PAH therapy as strata

5. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR) at Week 24
Description: PVR is a hemodynamic variable of pulmonary circulation and was measured by right heart catheterization (RHC). Per protocol, the change from baseline in PVR at Week 24 was reported for DBPC period.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of study treatment and who had a baseline measurement for the PVR.
Measure: Median (Full Range); unit: dynes*sec/cm^5
Arm/Group | Sotatercept Plus Background PAH Therapy (DBPC Period) | Placebo Plus Background PAH Therapy (DBPC Period)
Number analyzed (Participants) | 163 | 160
dynes*sec/cm^5 | -165.1 [-184.0 to -152.0] | 32.8 [24.0 to 40.0]
Statistical Analysis 1: Comparison: Sotatercept Plus Background PAH Therapy (DBPC Period) vs Placebo Plus Background PAH Therapy (DBPC Period); Test type: Other; p < 0.001, ARSW test — A 2-sided p-value was calculated using ARSW test with WHO FC II/III and background PAH therapy as strata; [statistical method as in outcome 1, analysis 1]; Treatment difference = -234.6, 95% CI 2-sided [-288.37 to -180.75] — Hodges-Lehmann location-shift estimate of the overall treatment difference with 95% CI was reported

6. Secondary Outcome: Change From Baseline in NT-proBNP Levels at Week 24
Description: NT-proBNP is a circulating biomarker that reflects myocardial stretch. Per protocol, the change from baseline in NT-proBNP level at Week 24 was reported for DBPC period.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of study treatment and who had a baseline measurement for the NT-proBNP levels.
Measure: Median (Full Range); unit: pg/mL
Groups:
- Placebo Plus Background PAH Therapy (DPBC Period): Participants received dose matched placebo SC injection every 21 days plus background PAH therapy during the DBPC period for up to approximately 24 weeks.
Arm/Group | Sotatercept Plus Background PAH Therapy (DBPC Period) | Placebo Plus Background PAH Therapy (DPBC Period)
Number analyzed (Participants) | 163 | 160
pg/mL | -230.3 [-236.0 to -223.0] | 58.6 [44.0 to 73.0]
Statistical Analysis 1: Comparison: Sotatercept Plus Background PAH Therapy (DBPC Period) vs Placebo Plus Background PAH Therapy (DPBC Period); Test type: Other; p < .001, ARSW test — A 2-sided p-value was calculated using ARSW test with WHO FC II/III and background PAH therapy as strata; [statistical method as in outcome 1, analysis 1]; Treatment difference = -441.6, 95% CI 2-sided [-573.54 to -309.61] — Hodges-Lehmann location-shift estimate of the overall treatment difference with 95% CI was reported

7. Secondary Outcome: Change From Baseline in the Percentage of Participants Who Improve in WHO FC at Week 24
Description: The severity of participant's pulmonary arterial hypertension (PAH) symptoms will be graded using the WHO FC system. WHO functional classification for PAH ranges from Class I (no limitation in physical activity, no dyspnea with normal activity), Class II (slight limitation of physical activity), Class III (marked limitation of physical activity) and Class IV (cannot perform a physical activity without any symptoms, dyspnea at rest). Participants who improve in WHO FC were classified into "Improved", "No change" and "Worsened". Improvement = reduction in FC, worsened = increase in FC and no change = no change in FC. Per protocol, change from baseline in the percentage of participants who improve in WHO FC at Week 24 were reported for DBPC period.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of study treatment and who had a baseline measurement for the WHO FC.
Measure: Number; unit: Percent change
Arm/Group | Sotatercept Plus Background PAH Therapy (DBPC Period) | Placebo Plus Background PAH Therapy (DBPC Period)
Number analyzed (Participants) | 163 | 159
Percent change | 29.4 | 13.8
Statistical Analysis 1: Comparison: Sotatercept Plus Background PAH Therapy (DBPC Period) vs Placebo Plus Background PAH Therapy (DBPC Period); Test type: Other — A 2-sided p-value was calculated using CMH method with WHO FC II/III and background PAH therapy as strata; p < 0.001, Cochran-Mantel-Haenszel

8. Secondary Outcome: Time to Death or the First Occurrence of Clinical Worsening Event
Description: Clinical Worsening events are defined as any of the following: worsening-related listing for lung and/or heart transplant; need to initiate rescue therapy with an approved background PAH therapy or the need to increase the dose of infusion prostacyclin by 10% or more; need for atrial septostomy; hospitalization for worsening of PAH (≥ 24 hours); or deterioration of PAH defined by both of the following events occurring at any time: worsened WHO FC and decrease in 6MWD by ≥15% confirmed by 2 tests at least 4 hours apart, but no more than 1 week. Per protocol, time to death or the first occurrence of clinical worsening event was reported.
Time Frame: Up to approximately 18 months
Population: All randomized participants who received at least one dose of study treatment and who died or experienced a first clinical worsening event.
Measure: Median (Standard Deviation); unit: Weeks
Arm/Group | Sotatercept Plus Background PAH Therapy | Placebo Plus Background PAH Therapy
Number analyzed (Participants) | 163 | 160
Weeks | NA (NA) — NA = Median time and standard deviation (SD) could not be calculated due to insufficient number of participants who had the first occurrence of clinical worsening event or died. | NA (NA) — NA = Median time and standard deviation (SD) could not be calculated due to insufficient number of participants who had the first occurrence of clinical worsening event or died.
Statistical Analysis 1: Comparison: Sotatercept Plus Background PAH Therapy vs Placebo Plus Background PAH Therapy; Test type: Other — A 2-sided p-value was calculated using Log rank test with WHO FC II/III and background PAH therapy as strata; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.163, 95% CI 2-sided [0.076 to 0.347] — Cox proportional hazard model was used to generate hazard ratio (HR) and 95% CI was reported with treatment group as the covariate stratified by the WHO FC II/III and background PAH therapy

9. Secondary Outcome: Change From Baseline in Percentage of Participants Who Maintain or Achieve a Low Risk Score Using the Simplified French Risk Score Calculator at Week 24
Description: The simplified French risk scoring system was based on the 2015 European Society of Cardiology (ESC)/European Respiratory Society (ERS) guidelines for the diagnosis and treatment of pulmonary hypertension (PH). In this study, the noninvasive parameters were used to determine the score. 'Low risk' was defined as attaining or maintaining all 3 low-risk criteria: WHO FC I or II, 6MWD > 440 m, and NT-proBNP <300 ng/L. Per protocol, change from baseline in percentage of participants who maintained or achieved a low risk score using the simplified French risk score calculator at Week 24 was reported for DBPC period.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of study treatment and who had a baseline measurement for the low risk score.
Measure: Number; unit: Percent Change
Arm/Group | Sotatercept Plus Background PAH Therapy (DBPC Period) | Placebo Plus Background PAH Therapy (DBPC Period)
Number analyzed (Participants) | 162 | 159
Percent Change | 39.5 | 18.2
Statistical Analysis 1: Comparison: Sotatercept Plus Background PAH Therapy (DBPC Period) vs Placebo Plus Background PAH Therapy (DBPC Period); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 4, analysis 1]

10. Secondary Outcome: Change From Baseline in the Physical Impacts Domain Score of Pulmonary Arterial Hypertension - Symptoms and Impact (PAH-SYMPACT®) at Week 24
Description: The PAH SYMPACT is a 23-item questionnaire to measure pulmonary arterial hypertension (PAH)-related symptoms and impact of PAH on daily life. The physical impact domain consists of walking slowly on a flat surface, walking quickly on a flat surface, walking uphill, carrying things, doing light indoor household chores, washing, or dressing oneself, and needing help from others. Participants were asked to recall and report on each item experienced in past 7 days. Score for each item ranges from 0 (not difficult at all) to 4 (extremely difficult). A domain score was calculated by summing the individual responses for each item and dividing by the number of impact items (range: 0=no physical impact to 4=severe physical impact). A higher score indicated more severe physical impact. Per protocol, change from baseline in the physical impacts domain score at Week 24 was reported for DBPC period.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of study treatment and who had a baseline physical impact domain score.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Sotatercept Plus Background PAH Therapy (DBPC Period) | Placebo Plus Background PAH Therapy (DBPC Period)
Number analyzed (Participants) | 163 | 160
Score on a scale | -0.13 [-0.15 to 0.00] | 0.01 [0.00 to 0.14]
Statistical Analysis 1: Comparison: Sotatercept Plus Background PAH Therapy (DBPC Period) vs Placebo Plus Background PAH Therapy (DBPC Period); Test type: Other; p = 0.010, ARSW test — A 2-sided p-value was calculated using ARSW test with WHO FC II/III and background PAH therapy as strata; [statistical method as in outcome 1, analysis 1]; Treatment difference = -0.26, 95% CI 2-sided [-0.490 to -0.040] — Hodges-Lehmann location-shift estimate of the overall treatment difference with 95% CI was reported

11. Secondary Outcome: Change From Baseline in the Cardiopulmonary Symptoms Domain Score of PAH-SYMPACT® at Week 24
Description: The PAH SYMPACT is a 23-item questionnaire to measure PAH-related symptoms and impact of PAH on daily life. The cardiopulmonary symptoms consist of shortness of breath, fatigue, lack of energy, swelling in the ankles or legs, swelling in the stomach area, and cough. Participants were asked to recall and report on each item experienced in past 7 days. Score for each item ranges from 0 (no symptom at all) to 4 (very severe symptoms). The mean individual symptom item score was determined for each of the 6 items and a domain score was calculated by summing the mean individual symptom item scores and dividing by the number of items (range: 0=no cardiopulmonary symptoms to 4=severe cardiopulmonary symptoms). A higher score indicated more severe symptoms experienced. Per protocol, change from baseline in the cardiopulmonary domain score at Week 24 was reported for DBPC period.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of study treatment and who had a baseline cardiopulmonary domain score.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Sotatercept Plus Background PAH Therapy (DBPC Period) | Placebo Plus Background PAH Therapy (DBPC Period)
Number analyzed (Participants) | 163 | 160
Score on a scale | -0.12 [-0.14 to -0.06] | -0.01 [-0.03 to 0.02]
Statistical Analysis 1: Comparison: Sotatercept Plus Background PAH Therapy (DBPC Period) vs Placebo Plus Background PAH Therapy (DBPC Period); Test type: Other; p = 0.028, ARSW test — A 2-sided p-value was calculated using ARSW test with WHO FC II/III and background PAH therapy as strata; [statistical method as in outcome 1, analysis 1]; Treatment difference = -0.13, 95% CI 2-sided [-0.256 to -0.014] — Hodges-Lehmann location-shift estimate of the overall treatment difference with 95% CI was reported

12. Secondary Outcome: Change From Baseline in the Cognitive/Emotional Impacts Domain Score of PAH-SYMPACT® at Week 24
Description: The PAH SYMPACT is a 23-item questionnaire to measure PAH-related symptoms and impact of PAH on daily life. The Cognitive/Emotional Impact domain consists of thinking clearly, feeling sad, feeling worried, and feeling frustrated. Participants were asked to recall and report on each item experienced in past 7 days. Score for each item ranges from 0 (not difficult at all) to 4 (extremely difficult). A domain score was calculated by summing the individual responses for each item and dividing by the number of impact items (range: 0=no cognitive/emotional impact to 4=severe cognitive/emotional impact). A higher score indicated more severe cognitive/emotional impact. Per protocol, change from baseline in the cognitive/emotional impacts domain score at Week 24 was reported for DBPC period.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of study treatment and who had a baseline cognitive/emotional impacts domain score.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Sotatercept Plus Background PAH Therapy (DBPC Period) | Placebo Plus Background PAH Therapy (DBPC Period)
Number analyzed (Participants) | 163 | 160
Score on a scale | 0.00 [0.00 to 0.00] | 0.000007 [0.00 to 0.0006]
Statistical Analysis 1: Comparison: Sotatercept Plus Background PAH Therapy (DBPC Period) vs Placebo Plus Background PAH Therapy (DBPC Period); Test type: Other; p = 0.156, ARSW test — A 2-sided p-value was calculated using ARSW test with WHO FC II/III and background PAH therapy as strata; [statistical method as in outcome 1, analysis 1]; Treatment difference = -0.16, 95% CI 2-sided [-0.399 to 0.084] — Hodges-Lehmann location-shift estimate of the overall treatment difference with 95% CI was reported

ADVERSE EVENTS:
Time Frame: Up to approximately 19 months
Description: All-cause mortality was reported on all randomized participants. Serious and non-serious adverse events were reported on all randomized participants who received at least one dose of study treatment.
Groups:
- Sotatercept Plus Background PAH Therapy (LTDB Period): Participants received sotatercept dose titrated up to 0.7mg/kg SC injection every 21 days plus background PAH therapy during the LTDB period for up to approximately 72 weeks.
- Placebo Plus Background PAH Therapy (LTDB Period): Participants received dose matched placebo SC injection every 21 days plus background PAH therapy during the LTDB period for up to approximately 72 weeks.
Arm/Group | Sotatercept Plus Background PAH Therapy (DBPC Period) | Placebo Plus Background PAH Therapy (DBPC Period) | Sotatercept Plus Background PAH Therapy (LTDB Period) | Placebo Plus Background PAH Therapy (LTDB Period)
All-Cause Mortality (participants affected / at risk) | 0/163 | 6/160 | 2/159 | 1/142
Serious Adverse Events (participants affected / at risk) | 23/163 | 36/160 | 26/158 | 14/142
Other Adverse Events (participants affected / at risk) | 111/163 | 88/160 | 82/158 | 50/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept Plus Background PAH Therapy (DBPC Period) (N=163) | Placebo Plus Background PAH Therapy (DBPC Period) (N=160) | Sotatercept Plus Background PAH Therapy (LTDB Period) (N=158) | Placebo Plus Background PAH Therapy (LTDB Period) (N=142)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular device occlusion (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device leakage (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device physical property issue (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Pulmonary artery aneurysm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept Plus Background PAH Therapy (DBPC Period) (N=163) | Placebo Plus Background PAH Therapy (DBPC Period) (N=160) | Sotatercept Plus Background PAH Therapy (LTDB Period) (N=158) | Placebo Plus Background PAH Therapy (LTDB Period) (N=142)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (9) | 3 (3) | 8 (9) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 20 (21) | 12 (13) | 6 (7) | 3 (4)
Nausea (Gastrointestinal disorders) | 17 (25) | 17 (26) | 8 (11) | 3 (5)
Fatigue (General disorders) | 17 (20) | 12 (12) | 10 (12) | 4 (4)
Injection site pain (General disorders) | 11 (12) | 10 (12) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 8 (10) | 10 (10) | 6 (7) | 3 (3)
COVID-19 (Infections and infestations) | 24 (25) | 19 (19) | 24 (24) | 21 (21)
Nasopharyngitis (Infections and infestations) | 7 (9) | 9 (10) | 4 (4) | 5 (5)
Urinary tract infection (Infections and infestations) | 5 (5) | 3 (4) | 8 (8) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (9) | 5 (5) | 6 (7) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 7 (7) | 9 (9) | 3 (3)
Dizziness (Nervous system disorders) | 17 (20) | 3 (4) | 6 (6) | 7 (7)
Headache (Nervous system disorders) | 33 (41) | 24 (30) | 9 (9) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 12 (15) | 2 (2) | 6 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 (24) | 3 (3) | 25 (36) | 1 (5)
Rash (Skin and subcutaneous tissue disorders) | 9 (10) | 4 (5) | 5 (6) | 2 (2)
Telangiectasia (Skin and subcutaneous tissue disorders) | 17 (21) | 5 (5) | 12 (16) | 2 (4)
Flushing (Vascular disorders) | 9 (10) | 3 (5) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT04576988/Prot_SAP_000.pdf